CLINICAL TRIAL: NCT04632563
Title: Prevalence of Musculoskeletal Symptoms in the Cambridge NIHR BioResource
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Principal Investigator, Professor Andrew McCaskie, Professor of Orthopaedic Surgery / Head of Department, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: A095310
Record Dates: First submitted 2020-11-11; First posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Musculoskeletal Diseases; Musculoskeletal Injury
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Member of BioResource: Any BioResource member who consents to take part in the study and completes the study questionnaire.
  Interventions: Other: Questionnaire including MSK-HQ (Musculoskeletal Health Questionnaire)

INTERVENTIONS:
Other: Questionnaire including MSK-HQ (Musculoskeletal Health Questionnaire) — A questionnaire regarding musculoskeletal past medical history and current symptoms.

SUMMARY:
Musculoskeletal diseases, such as osteoarthritis, represent a large proportion of the global burden of disease with hip and knee osteoarthritis alone being the 11th greatest cause of disease burden.

The purpose of this study is to determine the level of musculoskeletal symptoms in members of the Cambridge National Institute for Health Research (NIHR) BioResource and see if this is associated with their possession of genetic markers that have been identified as being associated with osteoarthritis.

This will allow us to determine the real level of musculoskeletal symptoms in this large cohort of volunteers and provide basic information that could be used to facilitate further musculoskeletal research in the NIHR BioResource population.

DETAILED DESCRIPTION:
All active members of the Cambridge NIHR BioResource will be approached.

They will be sent an email outlining the purpose of the study and asking that if they would like to take part to please complete the online questionnaire which will be linked to in the email.

For those individuals who agree to participate and complete the questionnaire, the Cambridge NIHR BioResource will provide the genetic marker information it already holds for specific markers that are known to be associated with osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Member of the NIHR BioResource
* Willing to consent to participate

Exclusion Criteria:

* Previous self-report of osteoarthritis on joining BioResource

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All members of the Cambridge NIHR BioResource
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
MSK Symptom Levels | 3 months
  Musculoskeletal Symptoms in respondents
Osteoarthritis genetic marker | 6 months
  Possession (or not) of specific genetic markers for osteoarthritis (obtained from information already held by the NIHR BioResource)

SECONDARY OUTCOMES:
MSK Cohort | 6 months
  Identification of those with particular musculoskeletal injuries and conditions for future studies

CONTACTS AND LOCATIONS:
Overall Officials: Andrew McCaskie, Principal Investigator — University of Cambridge

IPD SHARING:
Plan to Share IPD: No
Sharing of participant level data does not fall within the consent or ethical approval of the study.